CLINICAL TRIAL: NCT01677624
Title: A Multicenter, Open-label Study for E7040 in Japanese Subjects With Hypervascular Tumor and Subjects With Arteriovenous Malformation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7040-J081-301
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-01

CONDITIONS: Hypervascular Tumor and Arteriovenous Malformation
Keywords: Hypervascular tumor; arteriovenous malformation; arterial embolization
MeSH Terms: conditions — Arteriovenous Malformations

ARMS (1):
- E7040 (Experimental)
  Interventions: Device: E7040

INTERVENTIONS:
Device: E7040 — E7040 of optimal particle size (-300 um, 300-500 um, or 500-700 um to fit in a target vessel, target lesion, or embolized area) as transcatheter study device will be administered .

SUMMARY:
To evaluate the efficacy and safety of transcatheter arterial embolization with E7040 in Japanese subjects with hypervascular tumor or arteriovenous malformation

ELIGIBILITY:
Inclusion criteria:

1. Subjects who are subject to any of the following vascular embolization therapies

1. Subjects with hepatocellular carcinoma (HCC) who have deep stained early stage tumor confirmed by dynamic computerized tomography (CT) after bolus intravenous infusion of contrast media and have a typical finding of hypervascular tumor, and are not amenable to resection and local therapy, and meet any of the following (a) to (c).

   1. 1 lesion of >50 mm in diameter
   2. 2 or 3 lesions of >30 mm in at least one diameter
   3. 4 or more lesions
2. Metastatic hepatic cancer Subjects with metastatic hepatic cancer who have deep stained early stage tumor confirmed by dynamic CT after bolus intravenous infusion of contrast media and have a typical finding of hypervascular tumor but not amenable to resection, and whose primary lesion and extrahepatic lesion are controlled.
3. Hypervascular tumor other than metastatic hepatic cancer Subjects with deep stained early stage tumor confirmed by dynamic CT after bolus injection of contrast media and who have a typical finding of hypervascular tumor other than the liver (e.g., renal cell carcinoma, bone soft tissue sarcoma) and meets any of the following (a) to (b).

   1. Subjects applicable to pre-operative arterial embolization therapy to reduce tumor size or volume of bleeding for safer conduct of surgical resection or local therapy (e.g., radiofrequency ablation (RFA))
   2. Subjects in stable general condition and are applicable to pain control treatment
4. Arteriovenous malformation:

Subjects with arteriovenous malformation (except for central nervous system, heart, and lung) confirmed by dynamic CT but at a low risk of undesirable reflux into systemic circulation and with vessel malformation suitable for particle embolization in size

2. Subjects with Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0-2 (PS 0-1 for metastatic hepatic cancer)

3. No carry-over effect of prior therapy or adverse drug reactions which may influence the embolic effect of E7040, if having a history of prior therapy time elapsed from the end of prior therapy to the start of E7040 embolization therapy should be: Surgery: greater than or equal to 6 weeks Local therapy: greater than or equal to 4 weeks Embolization for non-target vessel: greater than or equal to 4 weeks

4. With a survival of greater than or equal to 12 months after the prior arterial embolization therapy using E7040

Exclusion criteria:

1. Subjects with clinical symptom or brain metastasis or cerebral encephalopathy requiring medical treatment
2. Suspected to have hepatocellular carcinoma (HCC) judging from clinical findings in patients with any disease other than HCC
3. Previously treated with arterial embolization therapy in target vessel
4. Previously treated with arterial embolization therapy in non-target vessel, resection in target organ, or local therapy (e.g., RFA) (except for HCC patient)
5. Subjects expected to have artery-pulmonary vein shunt or right-to-left shunt, or those with a possible risk of influx of embolized particles into the central nervous system.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shin Maeda, Study Director — Oncology Clinical Development Section Japan/Asia Clinical Research Product Creation Unit Eisai Product Creation Systems
Locations (10):
- Japan (10):
  - Hirosaki, Aomori
  - Chikushino-shi, Fukuoka
  - Kurume, Fukuoka
  - Nishinomiya, Hyōgo
  - Kanazawa, Ishikawa-ken
  - Kagoshima, Kagoshima-ken
  - Tsu, Mie-ken
  - Okayama, Okayama-ken
  - Chuo-ku, Tokyo
  - Minato-ku, Tokyo

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 'Insufficient response' = Insuf Resp
Groups:
- Device E7040: An optimal dose and size (100 to 300 μm, 300 to 500 μm, 500 to 700 μm) of microsphere that best matches the pathology (i.e., vascular target, vessel size, and target lesion) and the extent of embolization were carefully selected.
Period: Overall Study
Arm/Group | Device E7040
Started | 28
Completed | 27
Not Completed | 1
Not completed — Insuf Resp: intra-articular hemorrhage | 1

BASELINE CHARACTERISTICS:
Population: The analysis was performed using the Safety Analysis Set defined as all participants who received the embolization therapy with E7040 and had at least 1 evaluable safety data after the procedure.
Arm/Group | Device E7040
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.6 (12.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Success Rate of Embolization in the Target Vessel
Description: Embolization performance was graded per 1 of 4 levels: (1) complete embolization, 100% disappearance of contrast enhancement in the target vessel as evaluated by post-embolization digital subtraction angiography; (2) intensive embolization, ≥80% disappearance; (3) moderate embolization, ≥50% and <80% disappearance; (4) mild embolization, <50% disappearance. Success rate was obtained by calculating the percentage of complete embolization and intensive embolization cases. Embolization performance evaluated by both the Imaging Evaluation Committee and by the Investigator or Subinvestigator.
Time Frame: Day 1 (embolization) up to Day 30 after treatment
Population: The analysis was performed using Full Analysis Set defined as all participants who received embolization therapy with E7040 and had at least one evaluable efficacy data after the procedure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Device E7040
Number analyzed (Participants) | 28
Percentage of participants
  Imaging Evaluation Committee | 100 [87.6 to 100]
  Investigator or Subinvestigator | 96.4 [81.6 to 100]

2. Secondary Outcome: Success Rate for Operability of Embolization
Description: Operability and usability were evaluated by the Investigator on the basis of the sense of resistance when E7040 was injected, and how smoothly the microspheres could pass through the catheter. The evaluation criteria are very easy to use, easy to use, difficult to use, very difficult to use. Success rate was obtained by calculating the percentage of very easy to use and easy to use cases.
Time Frame: Day 1 (embolization) up to Day 30 after treatment
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Device E7040
Number analyzed (Participants) | 28
percentage of participants | 100 [87.6 to 100]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from the time of the procedure up to 30 days post procedure (if a surgery or local therapy was performed for the lesions where embolization was applied, AEs were collected up to that point).
Description: The analysis was performed using the Safety Analysis Set defined as all participants who received the embolization therapy with E7040 and had at least 1 evaluable safety data after the procedure.
Arm/Group | Device E7040
Serious Adverse Events (participants affected / at risk) | 2/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Device E7040 (N=28)
cholangitis (Hepatobiliary disorders) | 1
hepatic failure (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Device E7040 (N=28)
Post embolisation syndrome (Injury, poisoning and procedural complications) | 22
Lymphocyte count decreased (Investigations) | 9
Aspartate aminotransferase increased (Investigations) | 7
Alanine aminotransferase increased (Investigations) | 5
Blood bilirubin increased (Investigations) | 3
Blood creatinine increased (Investigations) | 3
Blood pressure increased (Investigations) | 3
Blood urea increased (Investigations) | 3
C-reactive protein increased (Investigations) | 3
Blood urine present (Investigations) | 3
Protein urine present (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 3
Blood albumin decreased (Investigations) | 2
Blood glucose increased (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 2
White blood cell count increased (Investigations) | 2
Constipation (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 6
Decreased appetite (Metabolism and nutrition disorders) | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Hepatic function abnormal (Hepatobiliary disorders) | 2
Headache (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 2
Pelvic pain (Reproductive system and breast disorders) | 4
Pyrexia (General disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other